CLINICAL TRIAL: NCT04926896
Title: Clinical Randomized Controlled Study on the Evaluation of Minimally Invasive Ilium Osteotomy and Its Bone Repairing Effect
Brief Title: Evaluation of Minimally Invasive Ilium Osteotomy and Its Bone Repairing Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: West China Hospital (Other); Werner Wicker Klinik (Network); Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-254
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Control Group

STUDY DESIGN:
Intervention Model Description: Experimental group:
  Minimally invasive bone harvesting surgery group.
  Control group:
  Traditional iliac crest bone harvesting surgery group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive bone harvesting surgery (Experimental): 1. .Applying routine approach in iliac crest bone harvesting surgery, make a 4cm long incision before or after the iliac crest, slice skin and subcutaneous tissue by layer., exposing the iliac crest ridge, outer plate and part of the iliac crest bone.
  2. Use the cortical bone opening device to open two bone holes with a diameter of 7.5 mm side by side in the iliac bone cortex ,place disposable battery-powered bone harvesting device for iliac crest bone harvesting operations.
  3. The direction of the tool bit should be parallel to the outer iliac plate, to avoid penetration of inner iliac layer, and avoid the injury to iliac blood vessels, nerves or internal organs.
  4. .Scrap and collect the cancellous bone by tool bit during operation.
  5. . After collecting sufficient amount of cancellous bone, turn off the power, screw out the cabin, and pour out the cancellous bone.
  6. . Suturing the iliac crest periosteum and deep fascia, closing the incision layer by layer, no drainage.
  Interventions: Procedure: Minimally invasive bone harvesting surgery
- Traditional iliac crest bone harvesting surgery (Placebo Comparator): 1. .Applying routine approach in iliac crest bone harvesting surgery, make a 4cm long incision before or after the iliac crest, slice skin and subcutaneous tissue by layer., exposing the iliac crest ridge, outer plate and part of the iliac crest bone.
  2. Use a bone chisel to open a lid on the iliac crest ridge cortex ,open the cover length at 3cm.
  3. Lift the iliac crest ridge cortex plate cover, use bone knife and scraper to harvest bone in the iliac bone marrow cavity.
  4. Avoid violence when using bone knives and scrapers, to avoid penetration of inner iliac layer, and avoid the injury to iliac blood vessels, nerves or internal organs.
  5. After collecting sufficient amount of cancellous bone, suturing the iliac crest periosteum and deep fascia, closing the incision layer by layer, no drainage
  Interventions: Procedure: Traditional iliac crest bone harvesting surgery

INTERVENTIONS:
Procedure: Traditional iliac crest bone harvesting surgery — The experimental group and the control group do not have special requirements; perform the surgery according to the normal operation methods of different sites.
  Arms: Traditional iliac crest bone harvesting surgery
Procedure: Minimally invasive bone harvesting surgery — Minimally invasive bone harvesting surgery
  Arms: Minimally invasive bone harvesting surgery

SUMMARY:
In this research, a new bone harvesting technique is introduced in order to find an iliac crest bone harvesting method for patients with less trauma, less postoperative pain in donor sites, and lower incidence of postoperative complications, so as to get ideal bone grafting materials at a small cost, enhance the effect of osteogenesis repair on bone defect or fusion site, and improve the operation quality.

DETAILED DESCRIPTION:
Based on the domestic and foreign research on minimally invasive bone harvesting, we have developed a disposable battery-powered bone harvesting device that can be used for milling bone tissues. Using this disposable battery-powered bone harvesting device, cancellous bone milling can be performed in a small bone hole with a diameter of 7.5 mm. The morselized bone or bone chips it milled can be used for bone fusion at the desired site. The technique adopts patented milling tool bit and electric drive, with high operation efficiency, so the surgery can be completed very quickly. The bone trauma in the operation can be significantly reduced and the pain in the donor site can be greatly alleviating. Moreover, the technique can obviously reduce the duration of bone harvesting and the cost of operating room. In addition, significant reductions in postoperative pain will also be helpful to a range of clinical advantages and benefits, such as the average hospitalization days, and will be expected to benefit significantly in patients undergoing autologous bone harvesting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinical bone defects or need for bone fusion;
2. Age 18 to 65, and gender is not limited;
3. Informed consent has been signed.

Exclusion Criteria:

1. Age less than 18 or greater than 65;
2. Patients with severe deformities of the iliac bone or extensive defects of the iliac bone, which are not suitable for bone extraction;
3. Patients with coagulation dysfunction;
4. Patients who are unwilling to perform iliac bone extraction;
5. BMI & lt; = 18.5 kg/m2;
6. Patients with type I and type II diabetes;
7. Osteoporosis(T & lt; = -2.5);
8. Moderate and severe anemia(hemoglobin & lt; 9g/L) or hypoproteinemia(albumin & lt; 30g/L);
9. Patients with malignant neoplasms; Patients with mental illness and those who are unconscious and unable to express themselves accurately.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2024-09-21 (Estimated); Study Completion 2024-12-21 (Estimated)

PRIMARY OUTCOMES:
the VAS score of pain in the donor site | 24 hours after the operation
  the VAS score of pain in the donor site
the comprehensive curative effect | 6 months after the operation
  the healing rate of the bone graft site

CONTACTS AND LOCATIONS:
Overall Officials: Yan Y Shigui, Professor, Study Director — Chief Scientist
Locations (1):
- Hangzhou Xinrun Medical Technology Co., Ltd., Hangzhou, Zhejiang, China